CLINICAL TRIAL: NCT05955027
Title: A Study to Evaluate the Effect of a Single Oral Dose of ZX-7101A on the QTc Interval in Healthy Subjects
Acronym: QTc-ZX-7101A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZX-7101A-206
Record Dates: First submitted 2023-06-14; First posted 2023-07-20 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational drug and the investigational drug placebo shall be provided by the sponsoring unit or its designated unit; Ensure that the placebo looks, tastes, and weighs similar to the test drug and marked for clinical trials; The test drug and placebo shall be blinded by the sponsor or its designated unit for each trial group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 80mg group (Experimental): D1, two 40mg tablets and two placebo tablets
  Interventions: Drug: ZX-7101A; Drug: Placebo
- 160mg group (Experimental): D1, four 40mg tablets
  Interventions: Drug: ZX-7101A
- Placebo group (Placebo Comparator): D1, 4 placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZX-7101A — a drug to treat influenza, oral
  Arms: 160mg group; 80mg group
Drug: Placebo — placebo control, oral
  Arms: 80mg group; Placebo group

SUMMARY:
The purpose of this study is to evaluate the effect of a single oral dose of ZX-7101A on the QTc interval in healthy subjects.

DETAILED DESCRIPTION:
Day 1, Oral fasting administration of ZX-7101A tablets 80mg, 160mg and placebo, 6 visit periods were set from days 2 to 15(Day2, Day3, Day5, Day7, Day10, Day15)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects, 18-45 years of age, inclusive, at the time of signing the ICF.
* Weight: Male weight ≥50 kg, female weight ≥45 kg, BMI between 19.0 and 28.0 kg/m2 (including cut-off value), BMI= weight (kg)/height 2 (m2).
* The investigator judged the subjects to be in good overall health based on their medical history, physical examination, vital signs, 12-lead electrocardiogram, laboratory tests (routine blood work, urine work, blood biochemistry, coagulation function), viral serology, and chest X-ray results (normal or abnormal test results have no clinical significance).
* Female subjects of childbearing potential and male subjects with a partner of childbearing potential who voluntarily signed ICF should be no fertile, sperm/egg donation for 6 months (female) or 90 days (male) from the beginning to the last dose, and voluntary use highly effective contraception (including partner) (non-drug contraception is required during the trial).
* Fully understand the trial content and possible adverse reactions, have the ability to communicate with researchers normally, while complying with study requirements, follow protocol procedures and restrictions, and be able to visit on time.

Exclusion Criteria:

* Subjects with a prior or present history of clinically abnormal metabolic, liver, kidney, hematological, pulmonary, cardiovascular, gastrointestinal, urinary, endocrine, neurological, or psychiatric disease who were judged by the investigator to be unsuitable for participation in this study.
* Subjects with digestive tract disease or any condition that may affect drug absorption, such as a history of liver and gallbladder disease, gastrointestinal disease, gastrointestinal surgery (except appendectomy) or a history of chronic pancreatitis, idiopathic acute pancreatitis, or habitual diarrhea.
* Subjects with electrolyte metabolism disorders such as hyperkalemia, hypokalemia, hypermagnesia, hypomagnesia, hypercalcemia or hypocalcemia.
* Subjects who have a history of other risk factors for tachycardia, or a family history of a first-degree relative (i.e. biological parent, sibling, or child) of short QT syndrome, long QT syndrome, or sudden unexplained death in young age (≤40 years).
* Allergic constitutions (such as allergies to two or more drugs, foods, and pollen), or determined by the investigator, may be allergic to the investigational product or any component of the investigational product.
* Subjects who have got acute respiratory infections within 2 weeks before screening; Or have a history of fungal infection.
* For patients with abnormal vital signs (blood pressure, pulse rate, ear temperature) and clinically significant results, the abnormal values of each vital sign are: Body temperature (ear temperature) >37.5 ℃; Systolic blood pressure (recumbent) <90 mmHg or ≥140 mmHg;Diastolic blood pressure (lying) <50 mmHg or ≥90 mmHg; Pulse rate (lying position) <50 beats/min or >100 beats/min.
* QTcF interval > 450ms or < 300 ms (Fridericia's correction), or QRS>120ms.
* Subjects who have abnormal liver function: alanyl aminotransferase (ALT) or aspartate aminotransferase (AST) higher than the upper limit of normal or serum total bilirubin (TBIL) greater than 1.5 times the upper limit of normal, who judged clinical significance by investigators.
* Subjects estimate glomerular filtration rate <90 mL/min/1.73 m2.
* Subjects virus serological test (hepatitis B virus surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, treponema pallidum specific antibody TPPA) positive results.
* Subjects with a history of drug abuse (morphine, dimethylene dioxyamphetamine, methamphetamine, THC, ketamine, cocaine) or who screened positive for drug abuse.
* Women who are pregnant or breastfeeding, or who test positive for blood pregnancy.
* Subjects who have used any P-gp or CYP inducer or inhibitor within 30 days before screening, or any prescription or Chinese herbal medicine within 4 weeks before the start of the trial, or over-the-counter or health care products (including polyvalent cations and metal supplements, etc.) within 2 weeks before the start of the trial; It should have a longer time interval if the elimination half-life is longer-at least 5 elimination half-lives for the drug.
* Subjects who consumed more than 14 units of alcohol per week in the 6 months prior before screening (1 unit of alcohol =360mL beer or 45mL spirits with 40% alcohol or 150mL wine) or had a positive alcohol breath test or could not abstain during the trial.
* Subjects who smoked more than 5 cigarettes per day in the 3 months prior before screening or habitually used nicotine-containing products or could not give up during the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-08 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
ΔΔQTc -Placebo-corrected, baseline-adjusted QTc interval (ΔΔQTc) | Day1, Day2, Day3, Day5, Day7, Day10, Day15
  Placebo-corrected, baseline-adjusted QTc interval (ΔΔQTc) at designed time after single oral administration of ZX-7101A tablets 80mg and 160mg in healthy Chinese adults. ΔΔQTc：The change of QTc interval from baseline value (ΔQTc) at each time point after administration was calculated, and then the difference of ΔQTc between the experimental group and the placebo group at each time point was calculated(ΔΔQTc).

SECONDARY OUTCOMES:
T wave | Day1, Day2, Day3, Day5, Day7, Day10, Day15
  T-wave morphology,or absence
PK parameters | Day1, Day2, Day3, Day5, Day7, Day10, Day15
  Cmax of prodrug ZX-7101A and active metabolite ZX-7101 (mother drug)
TEAE | Day1, Day2, Day3, Day5, Day7, Day10, Day15
  Rate of Treatment-Emergent Adverse Events(TEAE)
U wave | Day1, Day2, Day3, Day5, Day7, Day10, Day15
  U-wave presence and absence
PK parameters | Day1, Day2, Day3, Day5, Day7, Day10, Day15
  AUC0-t of prodrug ZX-7101A and active metabolite ZX-7101 (mother drug)
PK parameters | Day1, Day2, Day3, Day5, Day7, Day10, Day15
  AUCinf of prodrug ZX-7101A and active metabolite ZX-7101 (mother drug)
PK parameters | Day1, Day2, Day3, Day5, Day7, Day10, Day15
  Tmax of prodrug ZX-7101A and active metabolite ZX-7101 (mother drug)

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No